CLINICAL TRIAL: NCT00377624
Title: Sodium Hyaluronate for Treatment of Chronic Painful Shoulder With Limitation of Motion Due to Glenohumeral Joint Osteoarthritis, Rotator Cuff Tear and/or Primary or Secondary Adhesive Capsulitis
Brief Title: HUPS: Hyalgan Use in Painful Shoulder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_8229
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Osteoarthritis of Shoulder
MeSH Terms: interventions — Hyaluronic Acid

INTERVENTIONS:
Drug: sodium hyaluronate

SUMMARY:
Three-arm, parallel, double-blind, masked observer, randomized, PB-Saline controlled clinical trial. In order to avoid problems in the interpretation of the final results due to disparate enrollment from various centers, the number of patients enrolled per site will be the same per site. Study patients will be randomized to receive either 20 mg sodium hyaluronate, 3 i.a. sodium hyaluronate injections, followed by 2 PBSaline mock i.a. injections or 5 i.a. PB-Saline control injections. One investigator will administer the injection and the joint assessor will be blinded to the study. The anterior or posterior approach for the shoulder injection will be used.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

INCLUSION CRITERIA:

1. Patients with chronic shoulder pain with all of the following: of at least 6 months, but not greater than 5 years duration without clinically significant improvement in shoulder pain over the past one month, and present at least 50% of the days during the previous month.
2. Patients who have failed conventional therapy including but not limited to the following: NSAIDs; one or more i.a. or local peri-articular steroid injections and physiotherapy (a minimum of one month of previous physiotherapy treatment is required.
3. At screening, patients on chronic analgesic/anti-inflammatory medication should have a VAS pain score of >/= 30 mm and </= 90 mm indicating a lack of adequate and sustained response to previous and current therapies. At screening, patients not on chronic analgesic/anti-inflammatory medication should have a VAS pain score of >/= 40 mm and </= 90 mm. If bilateral shoulder pain is present, the investigator will use the more painful shoulder.
4. At baseline, after all analgesic/anti-inflammatory medications have been discontinued for 2 weeks, patients should have a VAS pain score of >/= 40 mm and </= 90 mm.
5. Patients with a limitation of shoulder motion in at least 1 direction at screening and baseline for the following active range of motions: Abduction with scapula fixed must be </= 80°; internal rotation in abduction must be ,/= 55°, and/or external rotation in abduction must be 180°. These limitations of shoulder motion are in comparison to normal expected ranges.
6. Patients with a retained active Range Of Motion ("ROM") >/= 30 percent in all directions at screening and baseline to rule out frozen shoulder. The ROM should be: >/= 30° for abduction with scapula fixed, >/= 30° external rotation, and >/= 20° for internal rotation.
7. Patients with at least one of the following conditions as examined and determined by Investigator: Osteoarthritis of the Glenohumeral Joint (OA), Rotator cuff tear (complete or partial), Adhesive capsulitis of the shoulder.
8. Patients who are able to complete efficacy measurement questionnaires.
9. Patients who are willing to discontinue all NSAIDs or other analgesic medication taken for their shoulder pain at least 2 weeks prior to baseline evaluation, with the exception of acetaminophen 500-1000 mg (1-2 tablets) q.i.d., p.r.n. (maximum 8 tablets or 4 grams per day) which would be sole rescue medication. Acetaminophen must not be taken within 24 hours of any visits or valuations. Patients must also be willing to abstain from any i.a. or peri-articular injections for the shoulder during the course of the trial, except for the assigned study product.

EXCLUSION CRITERIA

A. GENERAL MEDICAL CONDITIONS

1. Women of childbearing potential may not be entered if pregnant, nursing, or not using effective method of contraception until all follow-up procedures are complete.
2. Participation in an experimental drug/device study within the previous 30 days.
3. Prior history of any malignancy, with the exception of basal cell carcinoma of the skin treated more than 2 years ago, unless specific permission of the Sponsor is granted.
4. Significant bleeding diathesis.
5. Active liver disease, conjugated bilirubin, renal insufficiency, abnormal blood counts, or any clinically significant laboratory value, which the investigator feels, may affect the evaluation of the patient.

B. MUSCULOSKELETAL RELATED

1. Major injury including sports related injury to the shoulder within the past year.
2. Patients with chronic shoulder pain more than 5 years duration.
3. Any cervical spine disease that could confound the clinical assessment; chronic acromioclavicular disease, thoracic outlet syndrome, active epicondylitis, or symptomatic carpal tunnel disease, any musculoskeletal disease that could confound the diagnosis/evaluation of the painful shoulder, or any neurological etiology of the pain and any acute infection of the joint.
4. Surgery to the study joint within the previous 12 months.
5. Inflammatory arthropathy such as rheumatoid arthritis, lupus, psoriatic arthritis or Milwaukee shoulder.
6. Frozen shoulder involving either shoulder.
7. Patients with clinically significant shoulder pain improvement in the past month.
8. Gout or calcium pyrophosphate diseases involving the upper extremity that has flared within the previous 12 months.
9. Intra-articular or local peri-articular corticosteroid injections to the study joint or shoulder within the previous 3 months; or to any other joint within the previous month; or any oral corticosteroid within the previous month. Steroid inhalants are permitted if the patient has been on a stable regimen for the past month and remains on this regimen throughout the course of the trial. Low dose aspirin (325 mg or less) as an anti-thrombotic treatment is permitted if stable for one month prior to Screening and stable throughout the trial.
10. Patients who never received i.a. or peri-articular corticosteroid therapy for the signal shoulder. This includes patients with contraindication(s) to corticosteroids.
11. Intra-articular hyaluronan in the study joint within the previous 12 months. Use of glucosamine-or chondroitin sulfate-containing products unless at Screening the patient is on stable doses for at least 4 months and willing to remain on these stable doses throughout the course of the trial. Use of bisphosphonates unless at Screening the patient is on stable doses for the past month and willing to remain on these stable doses throughout the course of the trial.
12. Patients with shoulder X-ray findings of acute fractures, severe loss of bone density, a vascular necrosis and/or severe deformity.
13. Patients with documented evidence of clinically significant shoulder joint deformities.
14. If patients are receiving or performing physical therapy at screening, this physical therapy regimen must have been stable during the one-month preceding screening and remain stable throughout the course of the trial.
15. Patients with primary extra-articular shoulder syndromes in the absence of intra-articular disease such as uncomplicated impingement syndrome without limitation in ROM, bursitis and tendinitis without evidence of adhesive capsulitis.
16. Patients with Kellgren-Lawrence Stage IV osteoarthritis of the glenohumeral joint.
17. Any arthrogram of the signal joint within the past 3 months.

C. CONCOMITANT CONDITIONS, DISEASES, MEDICATIONS AND/OR CLINICAL HISTORY.

1. Patients with known allergies to acetaminophen, lidocaine, hyaluronan, or avian products.
2. Patients requiring chronic analgesia for any other condition (including chronic pain in the contralateral shoulder or another joint) that may interfere with the evaluations of the signal shoulder.
3. Patients with a recurrent medical history of severe allergic or immune-mediated reactions.
4. Patients with active infection of the skin in the vicinity of the potential injection site.
5. Patients taking any agent reported to have symptom relief for arthritis or be a disease/structure modifying drug.
6. Patients on concomitant therapy with anticoagulants.
7. Patients with any inter-current disease(s) or condition(s) that may interfere with the free use and evaluation of the affected shoulder for the 6-month course of the trial.
8. Patients with any inter-current chronic disease(s) or condition(s) that may predispose them to a high probability of interfering with the completion of the 6 month follow-up of the study such as peptic ulcer, liver disease, severe coronary disease, renal disease, cancer, pregnancy, alcoholism, drug abuse, mental state, or other clinically significant condition.
9. Patients participating in any clinical trial within one month of trial entry.
10. In the opinion of the clinical investigator a clinically significant abnormal laboratory test result(s) that may place the patient at a health risk, impact upon the study, or the patient's ability to complete the study.
11. Patients unable to legally comprehend the details and nature of the study.
12. Patients who - in the judgment of the clinician - are likely to violate the protocol regulations or unlikely to complete the study for any reason.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602
Dates: Start 2002-01; Study Completion 2004-09

PRIMARY OUTCOMES:
Improvement in shoulder pain on movement in previous 24 hours, based upon 100 mm VAS score up to 3 months after baseline for the 3 i.a. and 5 i.a. sodium hyaluronate injections compared to PB-Saline control

SECONDARY OUTCOMES:
Maintenance or improvement from baseline in shoulder pain on movement in previous 24 hours based upon 100 mm VAS score up to 6 months after baseline of
sodium hyaluronate treated patients compared to PB-Saline.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, MT, ASCP, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States